CLINICAL TRIAL: NCT05876520
Title: Clinical and Radiographic Assessment of Nano-Bioactive Glass Combined With I-PRF Scaffold in Vital Pulp Treatments in Mandibular Molars With Closed Apices: A Triple Blinded "Randomized Controlled Trial"
Brief Title: Clinical and Radiographic Assessment of Nano-Bioactive Glass Combined With I-PRF Scaffold in Vital Pulp Treatments in Mandibular Molars With Closed Apices
Acronym: I-PRF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noor Mohammed Kamal Eldeen Ahmed Mohmammed Sayed, Resident of Endodontics, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENDO-3-7-2
Record Dates: First submitted 2023-05-09; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Vital Pulp Treatment in Mature Permanent Teeth With Irreversible Pulpitis

STUDY DESIGN:
Intervention Model Description: Total Pulpotomy in mature permanent teeth treated with Nano-bioactive glass mixed with I-PRF
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Total pulpotomy with I-PRF only (Other): Total pulpotomy is done in mature permanent molars followed by I-prf application. Topped with BC putty for coronal seal, RMGI and restored with composite as final restoration
  Interventions: Procedure: Total pulpotomy with I-prf mixed with Nano-bioactive glass

INTERVENTIONS:
Procedure: Total pulpotomy with I-prf mixed with Nano-bioactive glass — Total pulpotomy is done in mature permanent molars followed by I-prf mixed with Nano-Bioactive glass application. Topped with BC putty for coronal seal, RMGI and restored with composite as final restoration

SUMMARY:
Clinical, Radiographic and pain assessment of Vital pulp treatment in patients suffering from irreversible pulpitis in mature permanent molars. Total pulpotomy is investigated using I-prf only vs I-prf mixed with Nano-bioactive glass.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Symptomatic irreversible pulpitis in mature mandibular molars only will be involved.
* Tooth should give positive response to cold test
* Haemostasias should be achieved after total pulpotomy
* The tooth is restorable and free from advanced periodontal disease, cracks and splits.
* Patients should be free from any systemic disease that may affect normal healing and predictable outcome.
* Patients who will agree to the consent and will commit to follow-up period.
* Patients with mature root apices
* Patients with no internal or external resorption and no periapical lesions
* Soft tissues around the tooth are normal with no swelling or sinus tract.

Exclusion Criteria:

* Patients with immature roots.
* Haemostasias after 10 minutes can not be controlled after total pulpotomy
* Patients with any systemic disease that may affect normal healing.
* Patients with periapical lesions or infections.
* Pregnant females.
* Patients who could/would not participate in a 6 months follow-up.
* Patients with fistula or swelling
* Patients with necrotic pulp.
* Patients with old age.

Ages: 14 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Clinical , Radiographic and Success rate | 6 month follow up
  Presence or absence of clinical signs and symptoms + Radiographic periapical assessment + success rate based on Radiographic findings

SECONDARY OUTCOMES:
Pain intensity | Within the first 24 hrs upto the 7th day
  VAS used to record daily pain intensity

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine Ahmed, Study Director — Vice Dean of Faculty of Dentistry Cairo University; Ahmed S. Elsheshtawy, Study Chair — Lecturer of Endodontics; Ayah Abdolwahab, Study Chair — Lecturer of Biomaterials; Noor K. Sayed, Principal Investigator — Resident of Endodontics
Locations (1):
- Noor Mohammed Kamal Eldeen, Cairo, Egypt